CLINICAL TRIAL: NCT06063421
Title: A Randomized Controlled Trial (RCT) to Compare Efficacy of Nicotine Replacement Therapy (NRT) Versus Electronic Cigarettes (EC) for Quitting Tobacco Smoking in Pakistan
Brief Title: Comparison of Nicotine Replacement Therapy and Electronic Cigarettes for Smoking Cessation in Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Strategic Health Research Limited (Network)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QUITS 3.1
Record Dates: First submitted 2023-09-04; First posted 2023-10-02 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation; Electronic Cigarette Use
Keywords: comparison of electronic cigarettes and NRT; electronic cigarettes versus NRT; electronic cigarettes; E-cigarettes; Nicotine Replacement Therapy (NRT); Electronic Nicotine delivery Systems (ENDS); EC; NRT; Quit smoking; smoking cessation; Tobacco cessation; Alternate Nicotine Delivery Systems (ANDS)
MeSH Terms: conditions — Smoking Cessation; Vaping; Tobacco Use Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, open label, parallel design RCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotine Replacement Therapy (NRT) (Active Comparator): The arm will comprise participants that receive NRT. The NRT used will be combination therapy; transdermal Nicotine patches will be combined with faster-acting oral products like gum or lozenges. The strength of nicotine patches will be from 7 to 21 mg, and for gum or lozenges, the strength will be 1-4 mg. Usage will be in the form of a daily nicotine patch and ad libitum use of the faster-acting lozenge to curb nicotine cravings. Participants will be provided with a 12-week supply of NRT.
  Interventions: Drug: Nicotine Replacement Therapy
- Electronic Cigarettes (EC) (Experimental): Participants randomised to the EC group will be supplied with an EC starter kit. The kit will consist of a personal vaping device with an integrated battery. Three commonly used flavours of e-liquid (tobacco, menthol, and fruit flavours) will be provided. All e-liquids will have a nicotine concentration of 18-20 mg/ml. EC will be provided for a total of 12 weeks.
  Interventions: Device: Electronic Cigarette (EC)

INTERVENTIONS:
Device: Electronic Cigarette (EC) — The intervention consists of the use of an Electronic cigarette device namely the Vaporesso Gen Air 40 Vape Kit. This is a complete kit including the EC device, integrated battery, refillable tank, charging cable, coil replacements and user manual. Three e-liquid flavours will be provided; tobacco, menthol and fruit flavour.
  Other Names: e-cigarettes; electronic nicotine delivery system (ENDS); Alternative nicotine delivery systems (ANDS); e-cigs
  Arms: Electronic Cigarettes (EC)
Drug: Nicotine Replacement Therapy — NRT will be in the form of combination therapy with a transdermal nicotine patch (7, 14, or 21mg) and an oral product: either gum or lozenge in 1, 2, or 4mg strength.
  Other Names: NRT
  Arms: Nicotine Replacement Therapy (NRT)

SUMMARY:
Smoking is prevalent in Pakistan, and a large proportion of the adult population smokes cigarettes or uses other forms of tobacco. Smoking cessation programmes are not well established, and the few centres that offer cessation, only provide basic support without stop-smoking medicines or other aids that can help people quit. Internationally approved stop-smoking treatments like nicotine replacement therapy (NRT) are available in larger cities, but they are very expensive. This makes it difficult for the general population to use NRT to aid in their desire to quit smoking. In the past few years, the use of electronic cigarettes (EC) has increased manifold. These devices are freely available and are offered in a wide variety of types and flavours. EC are also cheaper compared to NRT, which makes them affordable for most smokers. EC are not considered smoking cessation tools and are not used or recommended by cessation services. This study wants to compare EC with NRT to see which treatment is more successful in helping people quit smoking. The premise is that EC are more effective than NRT. The study also wants to determine the cost of using EC compared to that of NRT, when used for quitting smoking.

The study will have a total of 438 participants who will be assigned randomly (by chance) to two groups: NRT and EC. 219 participants will be provided with NRT, and 219 with EC. The participants will be adult smokers presenting at designated smoking cessation centres who are seeking help in quitting smoking. The main focus of the study is to see if EC are more successful than NRT in helping people quit smoking at the end of one year.

This research will provide useful information on the effectiveness and safety of EC and help develop a smoking cessation policy tailored to the population of Pakistan.

DETAILED DESCRIPTION:
Background:

The use of tobacco in its various forms remains the most common cause of preventable deaths in the world. Every year, 8 million people worldwide die of tobacco-related diseases. The highest burden (80%) is in underdeveloped and developing countries like Pakistan. Pakistan is a country with the fifth-highest burden of tobacco use in the world, with more than 15.6 million adult smokers. 21.9% of adult males and 3.4% of adult females are current cigarette smokers. In Pakistan, every year, around 160,000 lives are lost to tobacco use, and the impact on the economy is more than 1 billion dollars.

Despite this, smoking cessation services are not well established and are limited to a few facilities, predominantly in urban centres. These facilities don't have well-established cessation support programmes, and only provide basic behavioural support. Smoking cessation medicine like Nicotine replacement therapy (NRT) is available in Pakistan but very expensive. Over the past decade, the use of EC has increased in many countries around the world. Evidence suggests that current smokers use EC to reduce the number of cigarettes smoked per day, and ex-smokers use EC most commonly for cessation purposes and to prevent relapse. EC use in Pakistan has also become more common in the past few years. Electronic cigarettes are readily available and significantly cheaper than NRT. EC have great potential as stop-smoking aids; however, EC are not prescribed or recommended for this purpose in any of the smoking cessation centres. The purpose of this study is to evaluate the efficacy, safety, and cost-effectiveness of EC versus NRT for smoking cessation in the adult population of Pakistan.

Design:

The study is a pragmatic, parallel, open-label, randomized controlled trial of NRT with EC. Participants will be adult smokers who are willing to quit and have no preference for NRT or EC. 438 participants will be enrolled. A baseline assessment will be carried out to determine the demographic profile (age, sex, location, socioeconomic measures like income status, education, and employment. A detailed smoking history, including numbers of cigarettes smoked per day, history of quitting, quit attempts, past use of NRT, and past use of EC, will be reviewed. A complete medical examination by qualified clinicians will be conducted to determine eligibility for the study. Eligible participants will be randomly assigned to one of two treatment arms: EC or NRT, with 219 participants in each arm. The study will be conducted in 10 cessation clinics (SCC) across six districts of Pakistan. The NRT arm will be given a combination therapy of a nicotine patch and a faster-acting oral product of their choice (gum or lozenge). The EC arm will be provided with a refillable, 3rd generation EC device and a choice of 3 e-liquid flavours: tobacco, menthol, and fruit. Enough e-liquid will be provided to last until the next supply which will be after an interval of 4 weeks. Further supplies of e-liquids will be provided based on participants preferences. Both arms will be given supplies for 12 weeks and provided with standard behavioural support. The primary outcome measure is self-reported sustained smoking cessation at 52 weeks (one year). This will be verified by carbon Monoxide (CO) validation. A level of less than 8 ppm will be considered abstinent. Secondary outcome measures are CO-validated self-reported sustained abstinence at 24 weeks, self-reported 7-day point prevalence abstinence at 4, 24 and 52 weeks, change in the number of cigarettes smoked per day, time to relapse, and frequency and severity of adverse effects. An analysis of the average cost of treatment per participant will also be conducted.

The analysis for each outcome will use intention-to-treat (ITT) principles. For the primary analysis, the proportion of people who remain abstinent at 52 weeks (1 year) will be determined, and a comparison will be done between the NRT and the EC groups. Because the data variables are categorical, Chi-squared test will be used for significance testing. In our secondary analysis, we will examine time to relapse using Kaplan-Meier curves with Log Rank test for significance testing and Cox regression for Hazard Ratio analysis. We will compare the RCT groups using Chi-squared and logistic regression analyses for the proportion of participants that remained abstinent at 4 weeks and 24 weeks. Rates of adverse reactions will also be compared between arms using Chi-squared tests. The trial will include a cost comparison of total cost of ownership to see which method is the cheaper method, which can then be viewed in relation to their respective quit rates.

Discussion:

This will be the first randomized controlled trial comparing the effectiveness of NRT with EC in Pakistan. Pakistan does not have a national tobacco cessation policy or programme. No research has been conducted to determine the best options available for tobacco cessation in Pakistan. This study is important as it will provide an opportunity to develop Pakistan's first evidence-based smoking cessation policy, which can lead to the development of a comprehensive tobacco cessation programme.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older).
* Current-smokers presenting to a cessation clinic expressing a desire to quit smoking.
* Has capacity to consent.
* Can read and understand the instructions in Urdu and/or English and follow the study instructions and procedures.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Currently using EC or NRT products.
* Already enrolled in another similar study.
* Not willing to quit.
* Patients who have had a recent cardiovascular event like unstable angina, stroke or myocardial infarction in the past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Carbon Monoxide (CO) validated sustained abstinence at 52 weeks (1 year) | 52 weeks from Target Quit day (TQD).
  The primary outcome measure will be a biochemically (carbon monoxide) validated abstinence from smoking measured at 52 weeks (1 year) post target quit day.

SECONDARY OUTCOMES:
Biochemically verified sustained smoking abstinence at 24 weeks after the Target Quit Day | 24 weeks from Target Quit Day.
  This outcome measure will be a biochemically (Carbon Monoxide) validated abstinence of smoking measured at 24 weeks post target quit day.

OTHER OUTCOMES:
Self-reported 7-day point prevalence abstinence at 4, 24 and 52 weeks. | This self-reported 7-day point prevalence will be conducted at 4, 24 and 52 weeks post target quit day.
  This will consist of self reported abstinence of smoking "not a puff" in the 7 days leading to the measurement.
Adverse reactions | Adverse reactions will be recorded on 1, 4, 8, 24 and 52 weeks post TQD.
  Any adverse reactions or adverse events experienced by the participants.
Change in number of cigarettes smoked per day (CPD). | CPD will be measured at 1, 4, 8, 24 and 52 weeks post TQD.
  In those participants who are not abstinent, cigarettes smoked per day will be noted to determine if there has been any change in the mean number of CPD from the baseline.
Product satisfaction rating | This will be measured at 1, 4, 8, 24 and 52 weeks post TQD.
  Participants will be asked to rate their satisfaction with using an EC or NRT in comparison with cigarettes. Satisfaction will be measured on a scale (Product Satisfaction scale) from 1 to 5, with 1 being the lowest and 5 the highest satisfaction rating.
Intervention cost per participant | 12 weeks from Target Quit day.
  The average intervention cost per participant will be calculated. Each treatment has two components: behavioural support and cost of the smoking cessation aid. Behavioural cost is the same for both groups and will be provided by the cessation clinics. The trial will provide both NRT and EC for a period of 12 weeks. Total cost of both NRT and EC supplies will be determined. This will be divided by the total number of participants utilizing that treatment to get the average cost per participant. This will enable a comparison of the expenses for the cessation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar Malik, MPH, Principal Investigator — Head of Statistics
Locations (1):
- Health Research Consulting, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study will share IPD once the study has been completed and results published. All relevant data like study protocol, statistical analysis, consent form, etc will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 months after publication of study for a period of 5 years.